CLINICAL TRIAL: NCT03828019
Title: Adalimumab vs. Conventional Immunosuppression for Uveitis Trial
Acronym: ADVISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9196
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Uveitis
Keywords: Immunosuppression; Adalimumab; Antimetabolites; Calcineurin inhibitors; Corticosteroid sparing
MeSH Terms: conditions — Uveitis | interventions — Adalimumab; Azathioprine; Cyclosporine; Methotrexate; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Randomized treatment assignment with allocation ratio: 1:1 and two stratification variables: (1) number of immunosuppressive drug patient is on at time of enrollment (zero vs. one); (2) Initial dose of prednisone patient will be on in trial (<30 mg/day vs. ≥30 mg/day). The unit of randomization is the patient,
Masking Description: Unmasked treatment administration and outcome assessments (participants, study ophthalmologists, visual function examiners, and study coordinators are all unmasked). Masked assessment of baseline, 1-month, 3-month, and 6-month photographic images and optical coherence tomography (OCT) by the Reading Center (graders masked).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adalimumab (ADA) (Active Comparator): Adalimumab administered by subcutaneous injection at dosage and frequency specified below; total duration of treatment is 12 months.
  Adults (≥ 18 years of age) and adolescents ≥30 kg: 80 mg as initial dose; one week later by 40 mg then 40 mg every two weeks. Adolescents <30 kg: 40 mg as initial dose; one week later 20 mg then 20 mg every 2 weeks.
  Interventions: Biological: Adalimumab (ADA)
- Conventional immunosuppression (CON) (Active Comparator): Conventional immunosuppressive agent selected by study ophthalmologist at dose and frequency specified below;12 month treatment duration.
  Azathioprine: initially 2 mg/kg/day; max dose 200 mg/day. Methotrexate initially 15mg/wk; max dose 25 mg/wk. Mycophenolate initially 1 gm twice daily (BID); max dose1.5 gm BID. Cyclosporine (Sandimmune - dose 2.5 mg/kg BID and Neoral dose 2 mg/kg BID. Tacrolimus initially 1 mg BID; max dose 3 mg BID.
  Interventions: Drug: Conventional immunosuppression (CON)

INTERVENTIONS:
Biological: Adalimumab (ADA) — Adalimumab is a fully-human monoclonal antibody to TNF-α, which is approved by the U.S. FDA for the treatment of non-infectious intermediate, posterior, and panuveitides in adults and children 2 years of age and older.
  Other Names: Adalimumab, Humira
  Arms: Adalimumab (ADA)
Drug: Conventional immunosuppression (CON) — The study ophthalmologist will select amongst the permissible drugs (methotrexate, mycophenolate mofetil or azathioprine for antimetabolites; cyclosporine or tacrolimus for calcineurin inhibitors) taking into account the side effect profile of each drug with respect to subject's clinical situation.
  Other Names: Azathioprine, Imuran , Cyclosporine; Methotrexate, Rheumatrex; Mycophenolate, CellCept; Cyclosporine, Sandimmune, Neoral; Tacrolimus, Prograf
  Arms: Conventional immunosuppression (CON)

SUMMARY:
Non-infectious intermediate, posterior, and panuveitides are chronic, potentially-blinding diseases. Vision-threatening cases require long-term therapy with oral corticosteroids and immunosuppression. Based upon preliminary data, adalimumab, a fully-human, anti-tumor necrosis(TNF)-α monoclonal antibody, now US FDA-approved for uveitis treatment, may be a superior corticosteroid-sparing agent than conventional immunosuppressive drugs. The ADVISE Trial is multicenter randomized, parallel-treatment, comparative effectiveness trial comparing adalimumab to conventional (small molecule) immunosuppression for corticosteroid spring in the treatment of non-infectious, intermediate, posterior, and panuveitides.

DETAILED DESCRIPTION:
Abstract from protocol: The uveitides are a collection of diseases characterized by intraocular inflammation. Collectively, they are the 5th leading cause of blindness in the US, and the estimated cost of treating them is similar to that of treating diabetic retinopathy. Non-infectious intermediate, posterior, and panuveitides have the highest rates of visual loss and typically are treated with oral corticosteroids and immunosuppression. The Multicenter Uveitis Steroid Treatment (MUST) Trial (a randomized, comparative effectiveness trial, which compared 2 treatment paradigms for these diseases, systemic therapy with corticosteroids and immunosuppression vs. regional therapy [the fluocinolone acetonide implant]), and Follow-up Study demonstrated the superiority of the systemic approach to the regional ocular approach in terms of long-term visual outcomes with essentially no increase in systemic side effects in the systemic group. One key to systemic therapy's success was the use of systemic immunosuppression in 88% of participants, coupled with tapering the prednisone to <7.5 mg/day, a relatively safe dose. Non-alkylating agents are typically the first choice and the most often used are azathioprine, methotrexate, mycophenolate, cyclosporine, and tacrolimus. The alkylating agents, cyclophosphamide and chlorambucil, are used less often because of concerns about potential increased malignancy risk. Data from the Systemic Immunosuppressive Therapy for Eye Diseases (SITE) Cohort Study suggest that each of the conventional, non-alkylating agent immunosuppressive drugs is effective in controlling the inflammation while permitting tapering prednisone in ~40-55% of patients; hence combination therapy often is needed. Furthermore, minimizing the daily dose of prednisone is important, as the risk of cardiovascular disease and mortality increase with the cumulative dose of oral corticosteroids. In June 2016, the fully-human, anti-TNF-α monoclonal antibody, adalimumab, was approved by the US Food and Drug Administration (FDA) for the treatment of uveitis. Anti-TNF-α monoclonal antibody therapy has revolutionized the management of the rheumatic diseases largely due to its superior efficacy compared to conventional Disease Modifying Anti-Rheumatic Drugs. Data from VISUAL III, the extension of the two phase 3 trials that led to the FDA approval of adalimumab for the treatment of uveitis, suggest that adalimumab may be superior to conventional immunosuppression, as ~75% of participants had controlled inflammation with prednisone doses <5 mg/day. The ADalimumab Vs. conventional ImmunoSupprEssion for uveitis (ADVISE) Trial is a randomized, comparative effectiveness trial comparing adalimumab to conventional agent immunosuppression for patients with non-infectious, intermediate, posterior, and panuveitides. The primary outcome is the ability to successfully taper prednisone to <7.5 mg/day by 6 months after randomization while maintaining control of the inflammation. Secondary outcomes include prednisone discontinuation by 1 year, visual acuity, and complications of uveitis and its treatment.

ADVISE is being conducted under investigational new drug (IND) 132532. Adalimumab was FDA approved for the treatment of non-infectious intermediate, posterior, and panuveitides in adult patients in 2016 and in pediatric patients 2 years of age and older in 2018. In 2016, prior to the approval for pediatric patients, the FDA determined that use of adalimumab for the treatment of non-infectious intermediate, posterior, and panuveitides in adolescent patients in the ADVISE Trial does not increase risk for these patients as the drug is approved for treatment of pediatric patients for other indications. Although conventional immunosuppressive drugs are the standard approach and in widespread use, these drugs are not FDA approved for treatment of non-infectious intermediate, posterior, and panuveitides, and therefore an IND has been issued for this trial.

ELIGIBILITY:
Inclusion criteria

1. Age 13 years or older
2. Weight 30 kg (66 lbs) or greater
3. Active or recently active (≤ 60 days) non-infectious intermediate, posterior, or panuveitis
4. Prednisone indication meets one of the following:

   1. Active uveitis requiring one of the following i. Initiation of prednisone at dose greater than 7.5 mg/day ii. Increasing prednisone dose to greater than 7.5 mg/day iii. Currently receiving dose greater than 7.5 mg/day
   2. Inactive uveitis on current dose greater 7.5 mg/day
5. Initiation or addition of an immunosuppressive drug (i.e., a conventional immunosuppressive drug or adalimumab) is indicated
6. If currently receiving a conventional immunosuppressive drug, the drug and dose have been stable for at least 30 days
7. Patient able and willing to self-administer subcutaneous injections or have a qualified person available to administer subcutaneous injections
8. If posterior segment disease is present, ability to assess activity in at least one eye with uveitis
9. Visual acuity of light perception or better in at least one eye with uveitis

Exclusion criteria

1. Active tuberculosis or untreated latent tuberculosis (e.g., positive interferon-γ release assay [Interferon-gamma release assay (IGRA) test, such as Quantiferon-gold)
2. Untreated active hepatitis B or C infection
3. Any of the following baseline lab values

   1. White blood count <3500 cells per microliter
   2. Platelets <100,000 per microliter
   3. Hematocrit <30%
   4. aspartate aminotransferase (AST) or alanine transaminase (ALT) >1.5 times (X) upper limit normal value
   5. Serum creatinine >1.1 times (X) upper limit normal value
4. Behçet disease
5. Multiple sclerosis or other demyelinating disease
6. For patients with anterior/intermediate or intermediate uveitis without systemic disease, abnormal magnetic resonance imaging (MRI) of the brain consistent with demyelinating disease
7. Severe uncontrolled infection
8. Receipt of a live vaccine within past 30 days
9. Moderate to severe heart failure (NYHA class III/IV)
10. Active malignancy
11. Use of anti-TNF monoclonal antibody therapy within past 60 days
12. History of adalimumab intolerance or ineffectiveness
13. Hypersensitivity to any of the study treatments or their excipients
14. Current treatment with an alkylating agent
15. Current treatment with more than one immunosuppressive drug, not including oral corticosteroids
16. Shorter-acting regional corticosteroids administered within the past 30 days in any eye(s) with uveitis
17. Long-acting ocular corticosteroid implants, i.e., fluocinolone acetonide implant (e.g., Retisert®, Yutiq™, Iluvien®) placed within past 3 years unless uveitis is active in all eye(s) with an implant
18. Systemic disease that is sufficiently active such that it dictates therapy with systemic corticosteroids or immunosuppressive agents at the time of enrollment
19. Immunodeficiency disease for which immunosuppressive therapy would be contraindicated according to best medical judgment
20. Pregnancy or lactation
21. For persons of child-bearing potential or impregnating potential, unwillingness to use appropriate birth control (abstinence, combination barrier and spermicide, hormonal, or intrauterine device) for the next 18 months or plans to become a biological parent within the next 18 months.

    * In the United Kingdom (UK), use of combination barrier and spermicide alone does not meet birth control requirements.

    † UK female study participants must use highly effective methods of contraception.

    UK male study participants must use condoms for at least 6 months after the end of study treatment and their female partners of child-bearing potential are recommended to use highly effective contraception for the same duration. In addition, male participants should not donate semen during therapy or for 6 months following discontinuation of study treatment.
22. Medical problems or drug or alcohol dependence problems sufficient to prevent adherence to treatment and study procedures.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Jabs, MD MBA, Study Chair — CCTand Evidence Synthesis, JHU, Bloomberg School of Public Health
Locations (26):
- United States (19):
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Anne Bates Leach Eye Hospital, University of Miami Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - National Eye Institute, Bethesda, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - University of Michigan Health System, Kellogg Eye Center, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - MidAtlantic Retina, Wills Eye Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Retina, Nashville, Tennessee
  - Vanderbilt University Eye Institute, Nashville, Tennessee
  - Retinal Consultants of Texas, Bellaire, Texas
  - University of Utah, Moran Eye Center, Salt Lake City, Utah
  - University of Washington, Medicine Eye Institute, Seattle, Washington
- Australia (2):
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - University of Sydney, Sydney
- United Kingdom (5):
  - University Hospital Birmingham, Edgbaston, Birmingham
  - Bradford Teaching Hospital NHS Foundation Trust, Bradford
  - Cambridge University NHS Trust, Cambridge
  - University Hospitals of Leicester, Leicester
  - Moorfields Eye Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
A public use dataset corresponding to the primary manuscript and compliant with HIPAA regulations will be prepared within 1 year of completion of data collection. An encrypted data set containing de-identified data, a data dictionary and other study documentation (e.g. protocol and study manuals) will be provide after the data use agreement has been executed (see access criteria below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after completion of data collection, the data set will be available upon request .
Access Criteria: Requests for access to data will be reviewed by the Executive Committee to confirm oversight authority approval (e.g. institutional review board (IRB) approval) and a minimum standard of scientific merit. Once a request is approved, the investigator will be required to sign a data use agreement approved by the Johns Hopkins Bloomberg School of Public Health Office of Research Administration. An encrypted data set containing de-identified data, a data dictionary and other study documentation (e.g. protocol and study manuals) will be provide after the data use agreement has been executed.

REFERENCES:
- [Derived] Teabagy S, Wood E, Bilsbury E, Doherty S, Janardhana P, Lee DJ. Ocular immunosuppressive microenvironment and novel drug delivery for control of uveitis. Adv Drug Deliv Rev. 2023 Jul;198:114869. doi: 10.1016/j.addr.2023.114869. Epub 2023 May 10. PMID 37172782

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes with uveitis
Groups:
- Adalimumab (ADA): Adalimumab administered by subcutaneous injection at dosage and frequency specified below; total duration of treatment is 12 months.
  Adults (≥ 18 years of age) and adolescents ≥30 kg: 80 mg as initial dose; one week later by 40 mg then 40 mg every two weeks. Adolescents <30 kg: 40 mg as initial dose; one week later 20 mg then 20 mg every 2 weeks.
  Adalimumab (ADA): Adalimumab is a fully-human monoclonal antibody to tumor necrosis factor (TNF-α), which is approved by the U.S. FDA for the treatment of non-infectious intermediate, posterior, and panuveitides in adults and children 2 years of age and older.
- Conventional Immunosuppression (CIN): Conventional immunosuppressive agent selected by study ophthalmologist at dose and frequency specified below;12 month treatment duration.
  Azathioprine: initially 2 mg/kg/day; max dose 200 mg/day. Methotrexate initially 15mg/wk; max dose 25 mg/wk. Mycophenolate initially 1 gm twice a day (BID); max dose1.5 gm BID. Cyclosporine (Sandimmune - dose 2.5 mg/kg BID and Neoral dose 2 mg/kg BID. Tacrolimus initially 1 mg BID; max dose 3 mg BID.
  Conventional immunosuppression (CON): The study ophthalmologist will select amongst the permissible drugs (methotrexate, mycophenolate mofetil or azathioprine for antimetabolites; cyclosporine or tacrolimus for calcineurin inhibitors) taking into account the side effect profile of each drug with respect to subject's clinical situation.
Period: Overall Study
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CIN)
Started | 114; 214 Eyes with uveitis | 113; 220 Eyes with uveitis
Primary Outcome 6 Months | 112; 211 Eyes with uveitis | 105; 204 Eyes with uveitis
Completed | 109; 206 Eyes with uveitis | 98; 190 Eyes with uveitis
Not Completed | 5; 8 Eyes with uveitis | 15; 30 Eyes with uveitis
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Lost to Follow-up | 1 | 6
Not completed — Incarcerated | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes with uveitis
Groups:
- Adalimumab (ADA): Adalimumab administered by subcutaneous injection at dosage and frequency specified below; total duration of treatment is 12 months.
  Adults (≥ 18 years of age) and adolescents ≥30 kg: 80 mg as initial dose; one week later by 40 mg then 40 mg every two weeks. Adolescents <30 kg: 40 mg as initial dose; one week later 20 mg then 20 mg every 2 weeks.
  Adalimumab (ADA): Adalimumab is a fully-human monoclonal antibody to TNF-α, which is approved by the U.S. FDA for the treatment of non-infectious intermediate, posterior, and panuveitides in adults and children 2 years of age and older.
- Conventional Immunosuppression (CON): Conventional immunosuppressive agent selected by study ophthalmologist at dose and frequency specified below;12 month treatment duration.
  Azathioprine: initially 2 mg/kg/day; max dose 200 mg/day. Methotrexate initially 15mg/wk; max dose 25 mg/wk. Mycophenolate initially 1 gm BID; max dose1.5 gm BID. Cyclosporine (Sandimmune - dose 2.5 mg/kg BID and Neoral dose 2 mg/kg BID. Tacrolimus initially 1 mg BID; max dose 3 mg BID.
  Conventional immunosuppression (CON): The study ophthalmologist will select amongst the permissible drugs (methotrexate, mycophenolate mofetil or azathioprine for antimetabolites; cyclosporine or tacrolimus for calcineurin inhibitors) taking into account the side effect profile of each drug with respect to subject's clinical situation.
- Total: Total of all reporting groups
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON) | Total
Number analyzed (Participants) | 114 | 113 | 227
Number analyzed (Eyes with uveitis) | 214 | 220 | 434
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [34 to 55] | 44 [34 to 59] | 44 [34 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 78 | 153
  Male | 39 | 35 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 15 | 33
  Not Hispanic or Latino | 96 | 98 | 194
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 81 | 82 | 163
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 101 | 192
  United Kingdom | 9 | 3 | 12
  Australia | 14 | 9 | 23
Duration of uveitis at baseline [Median (Inter-Quartile Range); unit: years] | 0.9 [0.2 to 4.2] | 0.9 [0.3 to 3.6] | 0.9 [0.3 to 3.9]
Uveitis diagnostic class at baseline [Count of Participants; unit: Participants]
  Intermediate | 8 | 10 | 18
  Anterior and intermediate uveitis | 20 | 12 | 32
  Birdshot chorioretinitis | 23 | 26 | 49
  Multifocal choroiditis with panuveitis | 10 | 9 | 19
  Serpiginous choroiditis | 2 | 4 | 6
  Punctate inner choroiditis | 3 | 2 | 5
  Sympathetic ophthalmia | 2 | 2 | 4
  Vogt-Koyanagi-Harada disease early stage | 7 | 6 | 13
  Vogt-Koyanagi-Harada disease late stage | 1 | 4 | 5
  Isolated retinal vasculitis or panuveitis with retinal vasculitis | 28 | 23 | 51
  Isolated choroiditis or panuveitis with choroiditis | 10 | 15 | 25
NEI-VFQ-25 [Median (Inter-Quartile Range); unit: units on a scale] — National Eye Institute (NEI) Visual Function Questionnaire (VFQ) (NEI-VFQ-25) ranges from 0 to 100. Higher score is better visual functioning. Scores measure overall health, overall vision, difficulty with near-vision activities, pain or discomfort in or around the eyes, difficulty with distance activities, driving difficulties, limitations with peripheral and color vision, and limitations in social functioning, role limitations, dependency, and mental health symptoms related to vision.
  units on a scale | 72 [57 to 80] | 73 [61 to 81] | 73 [59 to 81]
EQ-5D health related quality of life [Median (Inter-Quartile Range); unit: units on a scale] — EuroQol Goup 5 Dimension questionnaire (EQ-5D) measures health related quality of life. The range is -0.11 to 1 where a score of 1 indicates best possible health state
  units on a scale | 0.93 [0.83 to 1.00] | 0.84 [0.83 to 1.00] | 0.85 [0.83 to 1.00]
Short-Form Health Survey- 36 item Physical component [Median (Inter-Quartile Range); unit: units on a scale] — Health related quality of life Physical component, range 1 - 100. Higher scores are better health
  units on a scale | 52 [44 to 57] | 54 [48 to 57] | 54 [48 to 57]
Short-Form Health Survey- 36 item Mental component [Median (Inter-Quartile Range); unit: units on a scale] — Range, 1 - 100. Higher scores indicate better mental health
  units on a scale | 53 [39 to 57] | 52 [43 to 57] | 52 [42 to 57]
Best Corrected Visual Acuity (BCVA) [Median (Inter-Quartile Range); unit: Standard letters EDTRS eye chart] — Participants' visual acuity was measured by certified examiners with best refractive correction in place. Participants were challenged with reading letters on lines of the standard ETDRS eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until no more meaningful readings could be made and were scored by how many letters could be correctly identified. More letters read is associated with higher visual acuity. (85 standard letters = 20/20 vision)
  Standard letters EDTRS eye chart | 81 [71 to 87] | 81 [74 to 86] | 81 [71 to 86]
Eye lens status [Count of Units; unit: Eyes with uveitis] — Indicates prior cataract surgery or presence of lens opacity
  Eyes with uveitis
    Eye is phakic ( natural lens) with no opacity | 102 | 87 | 189
    Eye is phakic (natural lens) with opacity/cataract | 76 | 89 | 165
    Eye is pseudophakic (Interocular lens placed) | 33 | 42 | 75
    Eye is aphakic (natural lens removed) | 3 | 2 | 5
Retinal thickness at the center subfield [Median (Inter-Quartile Range); unit: um] — Central subfield thickness as measured by OCT at a fundus photograph reading center. Values > 300 are indicative of macular edema.
  um | 255 [229 to 318] | 247 [219 to 282] | 252 [224 to 299]
Immunotherapy at baseline [Count of Participants; unit: Participants] — Whether a patient was not taking a immunosuppressive drug at baseline. Randomized to assure equal proportion in ADA and CID arms
  Participants
    On no immunotherapy at baseline | 90 | 88 | 178
    On one immunotherapy drug at baseline | 24 | 25 | 49
On corticosteroids greater than of equal to 30 mg at baseline [Count of Participants; unit: Participants] — Whether patient was on a dose of corticosteroid (e.g., prednisone) at a dose >= 30 mg/day at start of baseline visit
  Participants
    On less than 30 mg corticosteroids | 29 | 27 | 56
    On greater than or equal to 30 mg corticosteriods | 85 | 85 | 170
    missing steroid treatment data at BL | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Corticosteroid-sparing Treatment Success Within the First 6 Months After Randomization
Description: Corticosteroid-sparing success is defined as achieving inactive uveitis for two consecutive visits >= 28 days apart while on <= 7.5 mg/day of corticosteroids. Uveitis status (active vs inactive) is determined by the study ophthalmologist after reviewing the eye exam and imaging. Steroid dose and uveitis activity from visit months 6,8,10 and 12 were included in the analysis. Generalized estimating equations were used to fit logistic regression models to compare the cumulative proportion of corticosteroid sparing between the two treatment groups over time while accounting for correlation between replicate measurements on the same individual with an unstructured covariance matrix. Results were reported at 6 months (primary outcome) and 12 months (secondary outcome).
Time Frame: 6 months
Population: Participants with follow-up data through the 6 month visit or had an event (corticosteroid sparing success) before they were lost to follow-up
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of participants
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 112 | 105
Cumulative proportion of participants | 0.69 [0.60 to 0.77] | 0.54 [0.44 to 0.64]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); The sample size estimation: Adalimumab was estimated to be successful in 75% of patients. The overall success rate with conventional immunosuppression was estimated to be 51%. A sample size of 222 (111 per treatment group) provided 90% power to detect a difference in cumulative percent of 75% versus 51%; Test type: Superiority; p = 0.029, Regression, Logistic; Adjusted for the 2 stratification variables (initial prednisone dose and immunosuppression use at baseline); Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.06 to 3.25] — Estimated parameter is the Odds Ratios (ADA/CID). Result greater than 1 indicates ADA is superior in achieving successful corticosteroid sparing

2. Secondary Outcome: Corticosteroid-sparing Treatment Success Within the First 12 Months After Randomization
Description: as for outcome 1
Time Frame: 12 months
Population: Participants with follow-up data through the 12 month visit or had an event (corticosteroid sparing success) before they were lost to follow-up
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of participants
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 111 | 100
Cumulative proportion of participants | 0.86 [0.78 to 0.92] | 0.77 [0.67 to 0.84]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Generalized estimating equations were used to fit logistic regression models to compare the cumulative proportion of corticosteroid sparing between the two treatment groups over time while accounting for correlation between replicate measurements on the same individual with an unstructured covariance matrix. 2 stratification variables (initial prednisone dose and immunosuppression use at baseline) were included; Test type: Superiority; p = 0.072, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.94 to 3.86] — Odds ADA/ Odds CID

3. Secondary Outcome: Corticosteroid Discontinuation Success by 6 Months
Description: Corticosteroid discontinuation success is defined as achieving inactive uveitis for two consecutive visits >= 28 days apart after discontinuing corticosteroids. Uveitis status (active vs inactive) is determined by the study ophthalmologist after reviewing the eye exam and imaging. Steroid dose and uveitis activity from visit months 6,8,10 and 12 were included in the analysis. Generalized estimating equations were used to fit logistic regression models to compare the cumulative proportion of corticosteroid discontinuation between the two treatment groups over time while accounting for correlation between replicate measurements on the same individual with an unstructured covariance matrix. Results were reported at 6 months and 12 months.
Time Frame: 6 months
Population: Participants with follow-up through the 6 months visit or had an event (discontinued corticosteroids) before lost to follow-up
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of participants
Groups:
- Conventional Immunosuppression (CON): Conventional immunosuppressive agent selected by study ophthalmologist at dose and frequency specified below;12 month treatment duration.
  Azathioprine: initially 2 mg/kg/day; max dose 200 mg/day. Methotrexate initially 15mg/wk; max dose 25 mg/wk. Mycophenolate initially 1 gm twice daily (BID); max dose1.5 gm BID. Cyclosporine (Sandimmune - dose 2.5 mg/kg BID and Neoral dose 2 mg/kg BID. Tacrolimus initially 1 mg BID; max dose 3 mg BID.
  Conventional immunosuppression (CON): The study ophthalmologist will select amongst the permissible drugs (methotrexate, mycophenolate mofetil or azathioprine for antimetabolites; cyclosporine or tacrolimus for calcineurin inhibitors) taking into account the side effect profile of each drug with respect to subject's clinical situation.
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 112 | 105
Cumulative proportion of participants | 0.15 [0.09 to 0.24] | 0.11 [0.06 to 0.18]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.30, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.67 to 3.46] — Odds ratio is ADA/CID where value greater than 1 indicates ADA is superior for corticosteroid (prednisone) discontinuation

4. Secondary Outcome: Corticosteroid Discontinuation Success by 12 Months
Description: as for outcome 3
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of participants
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 109 | 98
Cumulative proportion of participants | 0.55 [0.45 to 0.64] | 0.40 [0.30 to 0.50]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Generalized estimating equations were used to fit logistic regression models to compare the cumulative proportion of corticosteroid discontinuation between the two treatment groups over time while accounting for correlation between replicate measurements on the same individual with an unstructured covariance matrix. 2 stratification variables (initial prednisone dose and immunosuppression use at baseline) were included; Test type: Superiority; p = 0.028, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.06 to 3.19] — Odds ADA/ Odds CID where value greater than 1 indicate greater corticosteroid sparing success in the ADA group

5. Secondary Outcome: Corticosteroid Exposure Over 12 Months
Description: Corticosteroid dose was collected at baseline and months 1,2,3,4,5,6,8,10, and 12. Mean corticosteroid dose per day was estimated with a negative binomial model at 12 months.
Time Frame: 12 months
Population: Participants with follow up treatment data
Measure: Mean (95% Confidence Interval); unit: mg/day of steroid use over 12 months
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
mg/day of steroid use over 12 months | 11.8 [10.5 to 13.2] | 13.8 [12.3 to 15.4]
Statistical Analysis 1: Comparison: Adalimumab (ADA); Test type: Superiority; p = 0.061, negative binomial model; Ratio of rate of steroid (mg/day ADA/CID = 0.86, 95% CI 2-sided [0.73 to 1.01] — Number greater than 1 would indicate rate of steroid use is higher in participants assigned to ADA

6. Secondary Outcome: Best Corrected Visual Acuity Change at 12 Months
Description: Mean change in best-corrected visual acuity from baseline to 12 months. Participants' visual acuity was measured by certified examiners with best refractive correction in place. Participants were challenged with reading letters on lines of the standard ETDRS eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until no more meaningful readings could be made and were scored by how many letters could be correctly identified. More letters read is associated with higher visual acuity (85 letters is 20/20 vision). Visual acuity data was collected at baseline and months 1,2,3,4,5,6,8,10, and 12 and estimated at 12 months with a mixed model.
Time Frame: 12 months
Population: All participants
Measure: Mean (95% Confidence Interval); unit: Standard letters ETDRS eye chart
Units Other Than Participants: Eyes with uveitis
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 114 | 113
Number analyzed (Eyes with uveitis) | 212 | 214
Standard letters ETDRS eye chart | 3.6 [1.3 to 5.8] | 3.2 [1.7 to 4.6]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Mixed effects models were used with a linear link. The fixed effects included initial steroid dose and immunosuppression use at baseline. Additional visit indicators (months 1-12) and corresponding treatment by visit interaction terms. An unstructured correlation was used to model repeated measurements by eye . A person-level random intercept was added to account for between-eye correlations; Test type: Superiority; p = 0.77, Mixed Models Analysis; Difference in mean change from BL = 0.4, 95% CI 2-sided [-2.3 to 3.1]

7. Secondary Outcome: Macular Edema Over 12 Months of Follow up
Description: Macular edema is defined as central retinal thickness greater than or equal to 300 micrometers as measured by a masked grader's review of OCT images. Greater retinal thickness is associated with poorer vision. Outcome measure is the odds ratio comparing macular edema at 12 months to baseline macular edema. Macular edema was measured at baseline and months 3, 6, and 12. The odds ratio at 12 months was estimated with a mixed model.
Time Frame: 12 months
Population: Participants with follow up retinal thickness data at enrollment and the 12 month visit
Measure: Number (95% Confidence Interval); unit: Odds ratio
Units Other Than Participants: Eyes with uveitis
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
Number analyzed (Eyes with uveitis) | 198 | 188
Odds ratio | 0.34 [0.23 to 0.51] | 0.63 [0.42 to 0.94]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Mixed effects models with a log link were used to assess treatment differences . The outcome measure was the odds ratio of having macular edema (OCT central subfield thickness > 300 um) at 12 months compared to baseline (BL). The treatment effect was the ratio of Odds ratios (ADA/CID) at 12 months. Values less than one indicate improvement in macular edema for the ADA treatment group relative to the CID group. Decrease in subfield thickness is good; Test type: Superiority; p = 0.028, Regression, Logistic; Ratio of odds ratios = 0.55, 95% CI 2-sided [0.31 to 0.94] — estimate is the ratio of odds ratios - OR ADA / OR CID. Value less than 1 indicates ADA is better at reducing macular edema

8. Secondary Outcome: Incidence of Infections at 12 Months
Description: Incidence of infections over 12 months of follow-up. Participants were asked about occurrences since the previous visit of infections requiring antibiotic or antiviral treatment. Data was collected at months 1,2,3,4,5,6,8,10, and 12. The rate of infections at 12 months was estimated with a negative binomial model.
Time Frame: 12 months
Population: Participants with follow up after the baseline visit
Measure: Number (95% Confidence Interval); unit: Number of infections per person year
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
Number of infections per person year | 0.40 [0.27 to 0.61] | 0.37 [0.24 to 0.57]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Test type: Superiority; p = 0.76, negative binomial model; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.61 to 1.98]

9. Secondary Outcome: Elevated Levels of AST or ALT (Hepatoxicity) by 12 Months.
Description: Cumulative percent of participants having elevated levels of aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than twice the upper level of normal by 12 months. Elevated levels of AST and ALT may indicate decline in liver function. Lab values of AST and ALT were measured at baseline and months 1,2,3,4,5,6,8,10, and 12 and the cumulative percent of participants with elevated lab values by 12 months was estimated by Kaplan Meier methods.
Time Frame: 12 months
Population: Participants with follow-up that did not have elevated levels of AST or ALT at baseline
Measure: Number (95% Confidence Interval); unit: Cumulative percent of participants
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 111 | 110
Cumulative percent of participants | 2 [0 to 5] | 10 [4 to 16]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); . Kaplan Meier techniques and Cox proportional hazards models were used to evaluate time to event outcomes; Test type: Superiority; p = 0.014, Regression, Cox; Cox Proportional Hazard = 0.16, 95% CI 2-sided [0.04 to 0.70]

10. Secondary Outcome: Elevated Creatine (Nephrotoxicity) by 12 Months
Description: Cumulative percent of participants having elevated creatine values (creatine greater than 30% above baseline or creatine > 1.5 mg/dL) by 12 months. Increases in creatine levels may indicate decreased kidney function. Lab values of creatine were measured at baseline and months 1,2,3,4,5,6,8,10, and 12 and the cumulative percent of participants with elevated creatine at 12 months was estimated by Kaplan Meier methods.
Time Frame: 12 months
Population: Participants with follow-up that did not have elevated creatine at the time of enrollment
Measure: Number (95% Confidence Interval); unit: Cumulative percent of participants
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 111 | 110
Cumulative percent of participants | 13 [6 to 18] | 14 [7 to 20]
Statistical Analysis 1: Comparison: Adalimumab (ADA); Test type: Superiority; p = 0.74, Regression, Cox; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.43 to 1.82]

11. Secondary Outcome: EQ-5D (Health Utility)
Description: The EQ-5D (EuroQol Group - 5 Dimension questionnaire) is a participant reported validated questionnaire that measures the patient's health status in five dimensions of health: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The range of questionnaire index scores is -0.59 to 1 where score of 1 indicates best possible health. The outcome measure is the odds of having EQ-5D score of 1 (perfect health) at 12 months compared to the odds of having EQ-5d score = 1 at the baseline visit. Participants completed the EQ-5D questionnaire at baseline and months 3, 6 and 12. General estimating equations with a log link were used to assess the odds ratio at 12 months.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
Odds ratio | 0.89 [0.60 to 1.32] | 1.17 [0.78 to 1.74]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Test type: Superiority; p = 0.35, Ratio of odds ratios; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.43 to 1.34] — Treatment comparison is the ratio of the odds ratios for each treatment group (ADA/CID) at 12 months. Values greater than one indicate greater improvement in health for the ADA treatment group relative to the CID group

12. Secondary Outcome: General Health-related Quality of Life -Physical Component (SF-36)
Description: Standard Form 36 item (SF-36) questionnaire is a validated participant reported measure of health related-quality of life.
  The physical component summary (PCS) is a score derived from the SF-36 that reflects a person's physical well-being.
  Range of scores is 0 to 100. Higher scores indicated better physical health. The minimally important clinical difference is 3-5 points.
  Outcome measure is the change in physical health score from baseline to 12 months. Participants completed the questionnaire at baseline and months 3, 6, and 12. The mean change from baseline at 12 months was estimated with a mixed model.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Difference in score on a scale
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
Difference in score on a scale | -0.29 [-2.01 to 1.42] | -1.68 [-3.27 to -0.08]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Test type: Superiority; p = 0.24, Mixed Models Analysis; Mean Difference (Net) = 1.39, 95% CI 2-sided [-0.95 to 3.73]

13. Secondary Outcome: Quality of Life Mental Health Component Standard Form 36 Item (SF-36)
Description: Standard Form 36 item (SF-36) questionnaire is a validated participant reported measure of health related-quality of life.
  The mental health component summary (MCS) is a score derived from the SF-36 that reflects a person's mental health and well-being. Range of scores is 0 to 100. Higher scores indicate better mental health. The minimally important clinical difference is 3-5 points. Outcome measure is the change in mental health score from baseline to 12 months. Participants completed the questionnaire at baseline and months 3, 6, and 12. The change from baseline at 12 months was estimated with a mixed model.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Difference in score on a scale
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
Difference in score on a scale | 1.56 [-0.55 to 3.67] | 0.97 [-1.19 to 3.13]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Net) = 0.59, 95% CI 2-sided [-2.43 to 3.61]

14. Secondary Outcome: Vision-related Quality of Life
Description: Vision-related quality of life was measured by the vision targeted subscale (excluding general health) from the National Eye Institute Visual Functioning Questionnaire 25 item (VFQ-25). The VFQ-25 is a validated, participant reported measure of the aspects of visual functioning that are most important for persons who have chronic eye diseases. Higher scores indicate better vision. Scores range from 0 to 100. Meaningful difference is 4-6 points. Participants completed the VFQ-25 at baseline and months 3, 6 and 12. The outcome is the change in VFQ-25 from baseline to 12 months estimated with a mixed model.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Difference in score on a scale
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 113 | 110
Difference in score on a scale | 6.7 [4.7 to 8.7] | 5.1 [2.9 to 7.3]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Net) = 1.6, 95% CI 2-sided [-1.4 to 4.6]

15. Secondary Outcome: Cataract Surgery at 12 Months
Description: Cumulative percent of uveitis eyes having cataract surgery by 12 months. Whether the patient had cataract surgery in the prior time period was determined at baseline and months 1,2,3,4,5,6,8,10,12 and the cumulative percent of eyes having cataract surgery by12 months was estimated by Kaplan-Meier methods.
Time Frame: 12 months
Population: Participants with phakic (no prior cataract surgery at baseline) eyes and follow up information
Measure: Number (95% Confidence Interval); unit: Cumulative percent of eyes
Units Other Than Participants: Eyes with uveitis
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
Number analyzed (Participants) | 96 | 91
Number analyzed (Eyes with uveitis) | 176 | 172
Cumulative percent of eyes | 2 [0 to 5] | 11 [4 to 17]
Statistical Analysis 1: Comparison: Adalimumab (ADA) vs Conventional Immunosuppression (CON); Test type: Superiority; p = 0.009, Regression, Cox; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.07 to 0.67]

ADVERSE EVENTS:
Time Frame: From enrollment through the 12 months visit (end of treatment) non-serious events were reported on the monthly or bimonthly case report form. Non serious events were analyzed by counting persons who ever reported the event over the 12 month study. Serious adverse events were reported by the clinical site as the event occurred or the site became aware of the event. Adverse event information was available only for participants (ADA N = 113, CID N= 110) who continued in the study past enrollment.
Description: Non serious adverse events were collected in both systemic and non-systemic forms. The events were collected systematically (check off list) by asking participants if they experienced any occurrence of a specific diagnosis, event, or side effect symptom on the case report form at each clinic visit. Non-systemic data was collected by asking if the patient experienced any other event or diagnosis. Serious adverse event collection was non systematic via an expediated serious adverse event form.
Arm/Group | Adalimumab (ADA) | Conventional Immunosuppression (CON)
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/110
Serious Adverse Events (participants affected / at risk) | 16/113 | 13/110
Other Adverse Events (participants affected / at risk) | 108/113 | 104/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (ADA) (N=113) | Conventional Immunosuppression (CON) (N=110)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) — Causing greater than 6 line (30 letter) loss of vision
Iris bombe (Eye disorders) | 1 (2) | 0 (0)
retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Uveitis glaucoma (Eye disorders) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 4 (4) | 0 (0) — Greater than 6 line (30 letter) loss of vision
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ocular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Miscarriage of partner (Social circumstances) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 2 (2)
Vitreous hemorrahage (Eye disorders) | 1 (1) | 1 (1)
Post cataract surgery vision loss (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Post cataract surgery vision loss of greater than 6 lines
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (ADA) (N=113) | Conventional Immunosuppression (CON) (N=110)
Epiretinal membrane (Eye disorders) | 17 | 20
Abdominal pain (Gastrointestinal disorders) | 46 | 48
mouth ulcer (Gastrointestinal disorders) | 21 | 23
Diahrrhea (Gastrointestinal disorders) | 42 | 46
Gingival swelling (Gastrointestinal disorders) | 23 | 24
Nausea (Gastrointestinal disorders) | 42 | 52
Vomiting (Gastrointestinal disorders) | 15 | 18
Fatigue (General disorders) | 76 | 87
Impaired healing (General disorders) | 28 | 44
Covid-19 infection (Infections and infestations) | 11 | 17
Upper respiratory infection (Infections and infestations) | 8 | 2
Appetite disorder (Metabolism and nutrition disorders) | 38 | 46
Fat redistribution (Metabolism and nutrition disorders) | 30 | 30
Fluid retension (Metabolism and nutrition disorders) | 46 | 51
Muscular weekness (Musculoskeletal and connective tissue disorders) | 44 | 53
Myalgia (Musculoskeletal and connective tissue disorders) | 77 | 84
Dizziness (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 76 | 78
Tremor (Nervous system disorders) | 43 | 60
Depression/anxiety (Psychiatric disorders) | 60 | 67
Insomnia (Psychiatric disorders) | 77 | 79
Easy bruising (Skin and subcutaneous tissue disorders) | 55 | 59
Acne (Skin and subcutaneous tissue disorders) | 32 | 36
Alopecia (Skin and subcutaneous tissue disorders) | 38 | 52
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 21 | 23
Rash (Skin and subcutaneous tissue disorders) | 34 | 32
Swelling face (Skin and subcutaneous tissue disorders) | 51 | 67
Gastric reflux disease (Gastrointestinal disorders) | 52 | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03828019/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03828019/SAP_001.pdf
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03828019/ICF_002.pdf